CLINICAL TRIAL: NCT01619020
Title: Gut Microbiota and Colonic Gene Expression: A Lignan Trial in Humans
Brief Title: FlaxFx, A Research Study of the Effects of Flaxseed Lignans on Colon Health
Acronym: FlaxFx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Texas A&M University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: FHCRC IR 7532
Record Dates: First submitted 2012-04-16; First posted 2012-06-14 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Healthy; Colon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flaxseed Lignans (Active Comparator): Capsules
  Interventions: Dietary Supplement: Flaxseed Lignans
- Placebo (Placebo Comparator): Capsules
  Interventions: Dietary Supplement: Flaxseed Lignans

INTERVENTIONS:
Dietary Supplement: Flaxseed Lignans — We will use a specially formulated dietary lignan supplement (Lignan Research Inc., San Diego, CA) as a source of lignans for the lignan challenge in the screening study and as a daily supplement in the intervention. It is a flaxseed extract that contains SDG (269 mg/g; 50 mg/capsule), pinoresinol diglucoside (160 mg/g), and lesser amounts of caffeic (50 mg/g), ferulic (40 mg/g) and coumaric acids (30 mg/g). Lignan capsules and placebo capsules will be prepared by Lignan Research, Inc., a well-established supplement company that follows GMP.

SUMMARY:
Colorectal (CRC) cancer is the third most common cancer in the United States and its incidence is rising in younger populations. Diet seems to affect risk for CRC.

Many parts of our diet are processed and modified by the microbes or bacteria in our gut. There are many different types of bacteria in our gut, each one of us has a "community" of different types and amounts of each type.

When we eat flaxseeds, certain types of bacteria will process them - producing compounds that can then affect our body. How much of these compounds are produced by each person depends on the "community" of bacteria in the gut.

Flaxseed and in certain nuts contain lignans, compounds that may have health benefits. Gut bacteria can convert the lignans into biologically active compounds that in animal models prevent the development of colon cancer. The investigators will study how these biologically active compounds affect colon cell-signaling pathways important to colorectal cancer risk.

Results from our study will bridge the current knowledge from animal studies and epidemiologic studies and may help to inform approaches for future CRC prevention.

DETAILED DESCRIPTION:
Part 1 (Screening):

Potential participants submit a screening questionnaire for eligibility. Eligible participants will come for an orientation for Part 1. If they consent the study coordinator will measure their height and weight and give them all the materials to do the activities for Part 1.

1. Stool sample
2. Days 1-3: take a lignan pill for three days
3. Day 3: 24-hour urine collection.

No all participants will be eligible for Part 2.

Part 2 (Trial):

Eligible participants will come for an orientation and consent.

Activities:

1. 3-day food record
2. Stool sample
3. Fasting blood draw.
4. Colon cleanse (at home). 2 months- no study activities Period 1,

1. Day 0: Stool sample 2. Day 0: 24-h urine collection 3. Take study capsule daily for 2 months. 4. Day 54: Stool sample 5. Day 54: 24-hour urine 6. Day 55: Fasting blood draw 7. Day 60 Sigmoidoscopy with biopsies 2 months- no study activities Period 2

1. Day 0: Stool sample
2. Day 0: 24-h urine collection
3. Take the other study capsule daily for 2 months.
4. Day 54: Stool sample
5. Day 54: 24-hour urine
6. Day 55: Fasting blood draw
7. Day 60 Sigmoidoscopy with biopsies

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking men and women
* ages 20-45 y
* don't eat a lot of vegetables

Exclusion Criteria:

* chronic medical illness, history of gastrointestinal disorders (e.g., ulcerative colitis, Crohn disease, celiac sprue, HNPCC, familial adenomatous polyposis, pancreatic disease, previous gastrointestinal resection, radiation or chemotherapy) and cancer (other than non-melanoma skin cancer);
* pregnancy or lactation;
* weight change greater than 4.5 kg within past year;
* oral or IV antibiotic use within the past 3 months;
* alcohol intake of >2 drinks/day (2 drinks being equivalent to 720 ml beer, 240 ml wine, or 90 ml spirits);
* dietary fiber intake >15 g/day;
* abnormal renal, liver or metabolic test results at baseline;
* inability to swallow pills;
* contraindications to sigmoidoscopy;
* regular use of prescription or over-the-counter medications, including oral contraceptives;
* known allergy to nuts, seeds and flaxseed;
* intention to relocate out of study area within next 12 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
mRNA expression in colonic mucosal tissue (stroma and epithelial) and exfoliated cells in individuals with low- or high-ENL excretion. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Lampe, PhD Rd, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- FHCRC, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lampe JW, Kim E, Levy L, Davidson LA, Goldsby JS, Miles FL, Navarro SL, Randolph TW, Zhao N, Ivanov I, Kaz AM, Damman C, Hockenbery DM, Hullar MAJ, Chapkin RS. Colonic mucosal and exfoliome transcriptomic profiling and fecal microbiome response to a flaxseed lignan extract intervention in humans. Am J Clin Nutr. 2019 Aug 1;110(2):377-390. doi: 10.1093/ajcn/nqy325. PMID 31175806